CLINICAL TRIAL: NCT05208437
Title: Shorten the Time Required to Correct the Arrival of Complete Oral Feeding in Premature Infants Whose Corrected Gestational Age Are Less Than 32 Weeks
Brief Title: Shorten the Time Required to Correct the Arrival of Complete Oral Feeding in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: [2021]394
Record Dates: First submitted 2021-12-30; First posted 2022-01-26 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-02

CONDITIONS: Premature Infants
Keywords: premature infants; oral feeding
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete oral feeding intervention group (Experimental): Premature infants will be assessed 12 times a day before feedings using the Feeding Preparation Scale. Feeding of premature infants using different interventions based on the results of the Feeding Preparation Scale.
  Interventions: Behavioral: Complete oral feeding intervention
- Routine nursing care group (Active Comparator): Pre-feeding assessments will be performed from premature infants corrected for gestational age at 34 weeks. If the baby's vital signs are stable, the method of oral feeding and then nasal feeding is used, and feeding 8 to 12 times a day until the baby reaches complete oral feeding. Routine nursing care is identical to the control group.
  Interventions: Behavioral: Routine nursing care group

INTERVENTIONS:
Behavioral: Complete oral feeding intervention — Premature infants will be assessed 12 times a day before feedings using the Feeding Preparation Scale by trained nurses. Assess the premature infants by using the Feeding Preparation Scale. If the premature infant does not meet the oral feeding standard, let the premature infant use the non-nutritive sucking for 3 minutes before the nasal feeding. If the premature infant meets the oral feeding standard, use the non-nutritive sucking for 3 minutes, and refer to the feeding schedule for the premature infant.
  Arms: Complete oral feeding intervention group
Behavioral: Routine nursing care group — Pre-feeding assessments will be performed from premature infants corrected for gestational age at 34 weeks. If the baby's vital signs are stable, the method of oral feeding and then nasal feeding is used, and feeding 8 to 12 times a day until the baby reaches complete oral feeding.
  Arms: Routine nursing care group

SUMMARY:
Non-nutritive sucking combined with a step-by-step oral feeding regimen shortens the total oral feeding cycle in premature infants

DETAILED DESCRIPTION:
In order to improve the feeding of premature infants <32 weeks of gestation, a complete oral feeding intervention program is provided for premature infants, which combined the evaluation of oral feeding readiness, the evaluation of oral feeding performance, non-nutritional sucking intervention and progressive feeding program. Premature infants will be assessed 12 times a day before feedings using the Feeding Preparation Scale.

Assess the premature infants by using the Feeding Preparation Scale. If the premature infant does not meet the oral feeding standard, let the premature infant use the non-nutritive sucking for 3 minutes before the nasal feeding; if the premature infant meets the oral feeding standard, use the non-nutritive sucking for 3 minutes, and refer to the feeding schedule for the premature infant. The whole intervention stops until the premature infant achieves the full oral feeding. Length of time required for complete oral feeding of premature infants is compared between the intervention group and the control group to evaluate the effect of the complete oral feeding intervention program on improving the feeding of premature infants <32 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <32w;
* Admit within 72 hours of birth;
* The guardian signs the informed consent;
* OI (oxygenation index >300)

Exclusion Criteria:

* Newborns with severe congenital malformations or various chromosomal diseases, genetic metabolic diseases, severe neurological diseases;
* Newborns who die during the study;
* Newborns who drop out of the study;
* Newborns who have NEC during hospitalization

Ages: 0 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Transition time from the initiation oral feeding to full oral feeding | During the procedure
  Transition time was defined as the days needed from introduction of oral feeding to obtain autonomous oral feeding when the nasogastric tube was removed and all the daily milk volume was taken from the bottle.
  time of complete oral feeding

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Hu, PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China